CLINICAL TRIAL: NCT05874388
Title: Characterisation of the Cognitive Profile of Patients Suffering From Friedreich's Ataxia
Acronym: CPCAF
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C22-77; 2023-A00290-45 (Registry Identifier: IDRCB)
Record Dates: First submitted 2023-02-07; First posted 2023-05-24 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Friedreich Ataxia
Keywords: FRATAXINE
MeSH Terms: conditions — Friedreich Ataxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Comprising subjects free of any motor or cognitive impairment, recruited from healthy relatives of patients (siblings, cousins, spouses) or for adults, among healthy people who are not related to the patients but who have been made aware of the existence of this research and who would meet the eligibility criteria and consent to participate in the study. The study will take place in a single session, during a health care consultation, during which the previously selected patients will take the tests included in the battery on a computer dedicated for the study. The total duration of the test is 45 minutes. No further visits will be necessary.
- Symptomatic participants: The study will involve a group of adolescents and adults symptomatic with FA with a confirmed molecular diagnosis, followed in the genetics department of the Necker Hospital. The study will take place in a single session, during a health care consultation, during which the previously selected patients will take the tests included in the battery on a computer dedicated for the study. The total duration of the test is 45 minutes. No further visits will be necessary. The validation of the results obtained will be determined by the correlation indices between the cognitive test scores used and the demographic variables and disease parameters considered, in particular the number of GAA triplet repeats in the allele of the FXN gene that contains the fewest repeats.

SUMMARY:
Friedreich's Ataxia (FA) Friedreich's Ataxia is a neurodegenerative disease caused by a homozygous expansion of the GAA triplet repeats of the frataxin gene (FXN). FA usually begins in childhood or adolescence. It affects both boys and girls. At the neurophysiological level, FA is characterised by neuronal loss affecting the dorsal root ganglia, spinal cord and cerebellum. At present, daily exercise is the only way to combat the disease. There is no cure for Friedreich's ataxia. Clinically, FA mainly combines balance, movement coordination, articulation (dysarthria) with cardiac involvement and sometimes diabetes . After a few years of evolution, walking is no longer possible. Recent data ; also indicate disturbances in information processing and cognitive functioning. In short, FA involves adolescents who progressively lose walking, writing and speech for some; however, each patient progresses differently with respect to the disease, and this is the case with respect to motor and cognitive symptoms.

DETAILED DESCRIPTION:
The role of behavioural and cognitive assessment in the clinical trial The effectiveness of a treatment is ultimately determined by the elimination of the physiological cause of the disease and the alleviation of the symptoms that patients suffer. However, new treatments rarely eliminate all causes and symptoms of the disease. As long as the effectiveness of a treatment is unknown, it is subtle changes in parameters that decide whether the approach taken is worth pursuing. For a clinical trial which is supposed to evaluate the effectiveness of a treatment for Friedreich's Ataxia, it is therefore necessary to evaluate subtle changes in the functioning of the motor and cognitive system induced by the treatment. For this reason, the project is assembling a battery of tests that quantify the most important aspects of motor, cognitive and speech function in patients with FA. These tests are designed with the specific needs of FA patients in mind, i.e. on the one hand, the tests assess functions that are particularly important in view of the symptoms of Friedreich's disease indicated in the scientific literature, and on the other hand, the psychometric characteristics of the tests are adapted to the general abilities of FA patients. In this respect, it is important to point out that the expansion of the GAA repetition in people with Friedreich's disease varies from 150 to 1,000 triples (compared to 7 to 25 in the rest of the population), and that this large variation in the genotype of FA patients could potentially influence the cognitive profile of the participants. Previous studies have suggested the relationship between the number of repeats of the GAA triplet of the FXN gene and performance in cognitive assessment tests. Specifically, while in FA patients both alleles of the FXN gene contain an unusually high number of GAA repeats, performance in cognitive tests would correlate with the number of GAA repeats in the allele that contains fewer such repeats. Using this test battery, we are therefore able to achieve our main objective, i.e. to characterise the cognitive profile of FA patients as a function of the number of GAA triplet repeats of the FXN gene. Specifically, the test battery will establish whether motor, executive and speech symptoms affect patients differently according to their particular genetic characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Patient group :

Patients aged 13 years or older Patients with FA confirmed by genetic study Compliant patients willing to undergo all tests Enrolled in a social security scheme or beneficiary of such a scheme

Control group :

Subjects aged 13 years or older Genetic characterisation to exclude the presence of alterations in the FXN gene No motor or cognitive impairment Compliant subjects willing to undergo all tests Membership in a social security scheme or beneficiary of such a scheme

Exclusion Criteria:

* Patient group :

Optic atrophy or decreased visual acuity Opposition of the patient, or of his parents if the patient is a minor, to participation in the study Non compliant patient according to the Investigator's opinion Person subject to a legal protection measure

Control group :

Alteration in the frataxin gene Optic atrophy or decreased visual acuity Opposition of the patient, or of his parents if the patient is a minor, to participation in the study Non-compliant patient in the opinion of the Investigator Person subject to a legal protection measure

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will involve two groups:
  * a group of adolescents and adults symptomatic with FA with a confirmed molecular diagnosis, followed in the genetics department of the Necker Hospital
  * a control group comprising subjects free of any motor or cognitive impairment, recruited from healthy relatives of patients (siblings, cousins, spouses) or for adults, among healthy people who are not related to the patients but who have been made aware of the existence of this research and who would meet the eligibility criteria and consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
characterization of the cognitive profile of patients suffering from Friedreich's Ataxia as a function of the number of GAA triplet repeats in the allele of the FXN gene that contains the least number of repeats. | through study completion, an average of 3 years
  Correlation of cognitive test scores

SECONDARY OUTCOMES:
Characterization of the motor profile of patients with Friedreich's Ataxia according to demographic variables and parameters related to the disease | through study completion, an average of 3 years
  Correlation of motor test scores with demographic variables demographic variables, disease parameters
Characterization of the executive profile of patients with Friedreich's Ataxia according to demographic variables and parameters related to the disease | through study completion, an average of 3 years
  Correlation of scores on tests of executive functions
Characterization of the speech production profile of patients with Friedreich's Ataxia according to demographic variables and parameters related to the disease | through study completion, an average of 3 years
  Correlation of speech production assessment test scores with demographic variables, disease-related parameters
To determine which dimensions of cognitive functioning are affected in patients with Friedreich's Ataxia and to verify the sensitivity of tests aimed at evaluating these dimensions to detect deficits in patients compared to healthy healthy subjects. | through study completion, an average of 3 years
  Comparison of motor test scores between patients and controls. Comparison of executive function test scores between patients and controls. Comparison of speech evaluation test scores between patients and controls.

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Funalot, Principal Investigator — APHP
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No